CLINICAL TRIAL: NCT02987621
Title: Can Transcranial Direct Current Stimulation Improve Ambulation and Fatigue Resistance in People With MS?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Thorsten Rudroff, Assistant Professor, Colorado State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-6856H
Record Dates: First submitted 2016-12-05; First posted 2016-12-09 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham first, wash out 7 days, then tDCS (Experimental): Separated by a minimum of 7 days from the sham treatment in a counterbalance order, all participants will perform leg muscle strength and fatigue testing once with tDCS stimulation.
  Leg muscle strength testing will be measured by performing a series of maximal effort knee extension, knee flexion, plantar/dorsi-flexion trials.
  Sham: Less than 0V of Transcranial Direct Current Stimulation tDCS: Less than 10V of Transcranial Direct Current Stimulation
  Interventions: Device: tDCS
- tDCS first, wash out 7 days, then Sham (Experimental): Separated by a minimum of 7 days from the sham treatment in a counterbalance order, all participants will perform leg muscle strength and fatigue testing once with tDCS stimulation.
  Leg muscle strength testing will be measured by performing a series of maximal effort knee extension, knee flexion, plantar/dorsi-flexion trials.
  Sham: Less than 0V of Transcranial Direct Current Stimulation tDCS: Less than 10V of Transcranial Direct Current Stimulation
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Less than 10V of Transcranial Direct Current Stimulation. Sham 0V of Transcranial Direct Current Stimulation.
  Other Names: The Travel Model v2.0 Advanced tDCS Kit; The Brian Simulator

SUMMARY:
In this project the investigators will be using non-invasive brain stimulation on people with multiple sclerosis (PwMS) to improve leg muscle function. Two groups of participants will be recruited. One group will perform strength testing with and without the brain stimulation. The second group of participants will perform a fatigue task, pulling against a wire at a low level of force, with and without the brain stimulation. This type of brain stimulation has been shown to transiently improve strength and fatigue measures in other populations, e.g. aged, Parkinson's, and improve cognitive abilities in people with multiple sclerosis. It is the investigator's hope that the increases in performance seen in other patient groups will also occur in people with multiple sclerosis. Future investigations will look to apply the non-invasive brain stimulation technique during physical rehabilitation to improve short and long term outcomes related to physical function.

ELIGIBILITY:
Inclusion Criteria:

* Medically diagnosed with MS
* Moderate disability (Patient Determined Disease Steps score 2-6)
* Self-reported differences in function between the legs (2-5 on a 1-5 scale)
* People with MS with physician clearance

Exclusion Criteria:

* A relapse of disease symptoms in the last 60 days
* A condition unrelated to MS that would exacerbate fatigue, such as anemia, hypothyroidism, shiftwork-related fatigue, B12 deficiency, major sleep disorder, or major depressive disorder
* Medical diagnosis or condition that makes participating in exercise training dangerous, such as major renal, pulmonary, hepatic, cardiac, gastrointestinal, HIV, cancer (other than treated basal cell cancer), other neurological disorders, or pregnancy
* History of heart attack or current diagnosis of cardiovascular disease
* History of seizure disorders (or on medications known to lower seizure threshold), hydrocephalus (buildup of fluid in the brain), or diabetes
* Alcohol dependence or abuse (>2 drinks/day), or present history (last six months) of drug abuse
* History of significant traumatic brain injury or hydrocephalus
* Pregnancy
* Recent hospitalization (within the last 3 months) or enforced bed rest/sedentary state.
* Presence of metal is present or implanted device or metal object that is not safe for TMS.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Health and Exercise Science, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham First, Seven Day Wash Out, Then tDCS; tDCS First, 7 Day Wash Out, Then Sham: Separated by a minimum of 7 days, participants will perform leg muscle strength and fatigue testing once with tDCS and once with Sham in a counterbalanced order.
  Leg muscle strength testing will be measured by performing a series of maximal effort knee extension, knee flexion, plantar/dorsi-flexion trials. Note: the 6 minute walk test was not conducted.
  The fatigue testing will be measured by time to fatigue with isometric contraction of the knee extensors.
  tDCS: Less than 10V of Transcranial Direct Current Stimulation
  Sham tDCS: Sham 0V of Transcranial Direct Current Stimulation
Period: Overall Study
Arm/Group | Sham First, Seven Day Wash Out, Then tDCS | tDCS First, 7 Day Wash Out, Then Sham
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Crossover study
Groups:
- All Study Participants: Separated by a minimum of 7 days, participants will perform leg muscle strength and fatigue testing once with tDCS and once with Sham in a counterbalanced order.
  Leg muscle strength testing will be measured by performing a series of maximal effort knee extension, knee flexion, plantar/dorsi-flexion trials. Note: the 6 minute walk test was not conducted.
  The fatigue testing will be measured by time to fatigue with isometric contraction of the knee extensors.
  tDCS: Less than 10V of Transcranial Direct Current Stimulation
  Sham tDCS: Sham 0V of Transcranial Direct Current Stimulation
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Leg Muscle Strength With and Without tDCS.
Description: Knee extensor strength will be tested with tDCS (less than 10V) and sham stimulation (0V). Participants performed maximal voluntary contractions (MVCs) with the knee extensors to objectively determine the weaker leg as more-affected, which was afterwards confirmed by the subject's self-report and used for the subsequent endurance task. This task consisted of a sustained isometric contraction at 15% MVC until volitional task termination and was immediately followed by a post MVC.
  During tDCS, stimulation intensity was ramped up to 2 mA, started 90 second prior to the task, and extended until task failure or a maximum stimulation length of 20 minutes. For Sham, the current was ramped up to 2 mA, but turned off after 30 seconds.
Time Frame: At session 1 and minimum of 7 days later
Population: Crossover design
Measure: Mean (Standard Error); unit: Newtons
Groups:
- All Study Participants: Participants will perform leg muscle strength testing with tDCS. On a separate day they will repeat the leg muscle strength testing with Sham stimulation.
  Leg strength testing will be measured by performing a series of maximal effort knee extension, knee flexion, plantar/dorsi-flexion trials. Furthermore, participants perform a 6 minute walk.
  tDCS: Less than 10V of Transcranial Direct Current Stimulation
  Sham tDCS: Sham 0V of Transcranial Direct Current Stimulation
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
Newtons
  tDCS Stimulation | 323 (15)
  Sham Stimulation | 330 (98)

2. Primary Outcome: Leg Muscle Endurance With and Without tDCS.
Description: Knee extensor endurance (fatigue) will be tested with tDCS (less than 10V) and sham stimulation (0V), as reported as time to failure.
  During tDCS, stimulation intensity was ramped up to 2 mA, started 90 second prior to the task, and extended until task failure or a maximum stimulation length of 20 minutes. For Sham, the current was ramped up to 2 mA, but turned off after 30 seconds.
Time Frame: At session 1 and minimum of 7 days later.
Population: Crossover design
Measure: Mean (Standard Error); unit: seconds
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
seconds
  tDCS Stimulation | 1087 (938)
  Sham Stimulation | 872 (547)

3. Primary Outcome: 6 Minute Walk Test
Description: After completion of the tDCS/Sham strength assessment participants will perform a 6 minute walk test. The test will be performed in a cordoned off hallway with 2 cones placed 30 meters apart. Once the participants begin walking, a timer will be started and the distance covered every min will be recorded. Participants are allowed to stop and rest during the test if required. Every minute during the walk test participants will be asked their rating of perceived exertion (RPE, 0-10 scale).
Time Frame: At session 1 and minimum of 7 days later
Population: No data was collected
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were determined at session 1 and minimum of 7 days later at session 2. No adverse events were reported by participants.
Description: The six minute walk test was not performed and therefore no participants were at risk.
Groups:
- All Study Participants-Leg Muscle Strength tDCS: Knee extensor strength was tested for all study participants with tDCS (less than 10V). All study participants performed maximal voluntary contractions (MVCs) with the knee extensors to objectively determine the weaker leg as more-affected, which was afterwards confirmed by the subject's self-report and used for the subsequent endurance task. This task consisted of a sustained isometric contraction at 15% MVC until volitional task termination and was immediately followed by a post MVC.
  During tDCS, stimulation intensity was ramped up to 2 mA, started 90 second prior to the task, and extended until task failure or a maximum stimulation length of 20 minutes.
- All Study Participants-Leg Muscle Strength Sham: Knee extensor strength was tested for all study participants with sham stimulation (0V). All study participants performed maximal voluntary contractions (MVCs) with the knee extensors to objectively determine the weaker leg as more-affected, which was afterwards confirmed by the subject's self-report and used for the subsequent endurance task. This task consisted of a sustained isometric contraction at 15% MVC until volitional task termination and was immediately followed by a post MVC.
  For Sham, the current was ramped up to 2 mA, but turned off after 30 seconds and extended until task failure or a maximum length of 20 minutes.
- All Study Participants-Leg Muscle Endurance tDCS: Knee extensor endurance (fatigue) was tested for all participants with tDCS (less than 10V) as reported as time to failure.
  During tDCS, stimulation intensity was ramped up to 2 mA, started 90 second prior to the task, and extended until task failure or a maximum stimulation length of 20 minutes.
- All Study Participants-Leg Muscle Endurance Sham: Knee extensor endurance (fatigue) was tested for all participants with sham stimulation (0V) as reported as time to failure.
  The current was ramped up to 2 mA, but turned off after 30 seconds until task failure or a maximum length of 20 minutes.
Arm/Group | All Study Participants-Leg Muscle Strength tDCS | All Study Participants-Leg Muscle Strength Sham | All Study Participants-Leg Muscle Endurance tDCS | All Study Participants-Leg Muscle Endurance Sham
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT02987621/Prot_SAP_ICF_000.pdf